CLINICAL TRIAL: NCT06131359
Title: Pilot Study to Develop Protocols for Recording Electromyography Signals From Tibialis Posterior and Demonstrate Age-related Changes in Muscle Activity Which May be Linked to Tibialis Posterior Tendon Dysfunction (TPTD)
Brief Title: Pilot Study to Develop Protocols for Recording Tibialis Posterior EMG
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Robert Jones and Agnes Hunt Orthopaedic and District NHS Trust (Other Government)
Collaborators: University of Exeter (Other)
Responsible Party: Sponsor
Other Study IDs: RL1880
Record Dates: First submitted 2023-08-09; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Tibialis Posterior Dysfunction; Emg
Keywords: tibialis posterior; EMG; gait lab
MeSH Terms: conditions — Posterior Tibial Tendon Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Younger adults: age 18-35 years
  Interventions: Diagnostic Test: Fine wire EMG and Force Frame muscle strength testing
- Older adults: age over 55 years
  Interventions: Diagnostic Test: Fine wire EMG and Force Frame muscle strength testing

INTERVENTIONS:
Diagnostic Test: Fine wire EMG and Force Frame muscle strength testing — Insertion of fine wires for EMG study of tibialis posterior and assessment of muscle strength using a force frame

SUMMARY:
This is an observational pilot study to allow us to create a normal database of muscle function of one of the muscles in the back of the leg (tibialis posterior). Individuals with no foot and ankle problems will be recruited to undergo 2 tests.

Firstly, under ultrasound guidance we will insert a very fine needle into the muscle which is deep inside the lower leg. The needle is similar to an acupuncture needle and is removed once it is in the muscle. This leave behind 2 very fine wires (the size of strand of hair) which we will use to assess the electrical activity of the muscle when walking.

Secondly, we will test muscle strength by asking individuals to push against the side of a special box, called a force frame). This will give us a link between the muscle activity and the strength of the muscle.

We plan to recruit 30 individuals, (15 in each age group), 20 of whom will undergo repeat testing on a separate day to ensure our protocol is repeatable.

DETAILED DESCRIPTION:
Tibialis posterior (TP), plays a substantial role in supporting the arch of the foot. Tibialis posterior tendon dysfunction (TPTD) involves pain and swelling on the inner side of the foot and often leads to an acquired flat foot deformity. However, there is also a tendency for foot width to increase and arch height to decrease with age. Greater concurrent activation of muscles that perform opposing movements has been shown with age. However it is unknown whether greater co-activation of TP and its opposing peroneal muscles increase with age. There is uncertainty regarding the management of TPTD, recently highlighted by the James Lind Alliance as a research priority.

To improve understanding of TP function we can study the electrical signal when TP activates using electromyography (EMG). Foot arch height has been shown to influence the pattern of TP activation in young-middle aged adults during walking. However, to enable comparisons between groups of participants (e.g. young vs. old, or patients vs. healthy controls) it is necessary to perform a normalization process to account for individual differences e.g. in orientation of muscle fibres. Recent expert consensus advocated normalising to a maximum voluntary contraction (MVC) when comparing groups. Previous studies have reported poor between-day reliability of TP EMG when normalising to an MVC. In the latter studies, the MVC contraction was performed against manual resistance, potentially reducing the reliability of the measurement due to variability in the resistance from the tester. Reliability of the MVC may be improved by using a controlled means of providing resistance to muscle contraction such as an isokinetic dynamometer, or a ForceFrame (VALD Health). Establishing a reliable method to record EMG from TP will enable future work investigating the mechanisms leading to TPTD and explore the potential for EMG to tailor treatment plans.

Due to the depth of TP, it is necessary to use fine-wire electrodes, inserted under the skin to record EMG. Fine-wire insertions will be performed by trained co-worker Dr Jo Reeves using ultrasound guidance and verified with electrical stimulation. Surface sensors will be placed on additional muscles (peroneals, tibialis anterior and gastrocnemii). With the electrodes in place the participants will lie on their backs and perform three maximum contractions of ankle inversion against resistance. The EMG signal from the contraction with the highest force value will be used to normalise subsequent EMG during walking. Participants will perform six walks on a standard walkway.

A target of 30 participants will be recruited (15 younger adults and 15 older adults). A subset of 20 participants will repeat the above procedure in a second session, separated by at least a day. Previous work on the between-day reliability of EMG recording from soleus during walking demonstrated comparable reliability using fine-wire electrodes to surface electrodes with 18 participants (Bogey et al., 2003). Reliability will be established with the standard error of measurement, the coefficient of variation, the intra-class correlation coefficient and the coefficient of multiple correlation.

ELIGIBILITY:
Inclusion Criteria:

* Adults will be included for the younger group if 18-35 years of age and the older group over 55 years of age.

Exclusion Criteria:

* Any recent lower limb injury or foot or ankle pathology including hallux valgus and tibialis posterior tendon dysfunction.
* Any cardiovascular, musculoskeletal or neurological conditions or disease, immune deficiency or haemophilia.
* Taking anti- biotic medication, anti-coagulant medication, and anti -platelet therapy.
* Walk with an aid.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Typically developing adult subjects
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
EMG signal amplitude and time profile across the gait cycle when walking | Baseline (and repeat on different day within 1 month for subgroup)
  Using fine wire
Muscle strength | Baseline (and repeat on different day within 1 month for subgroup)
  Using force frame

CONTACTS AND LOCATIONS:
Overall Officials: Catriona Heaver, Study Chair — RJAH; Caroline Stewart, Principal Investigator — RJAH; Jo Reeves, Principal Investigator — University of Exeter